CLINICAL TRIAL: NCT06852898
Title: Manual Therapy With Radial Extracorporeal Shockwave Therapy (ESWT) Compared to Manual Therapy Alone for the Treatment of Acute Mechanical Low Back Pain: A Randomized Clinical Trial
Brief Title: Comparative Clinical Trial: Manual Therapy With and Without Radial Extracorporeal Shockwave Therapy to Treat Acute Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeast College of Health Sciences (Other)
Responsible Party: Principal Investigator, Jeanmarie R. Burke, PhD, Dean of Faculty and Research, Northeast College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-08
Record Dates: First submitted 2025-02-17; First posted 2025-02-28 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Lower Back Pain
Keywords: chiropractic care; acute low back pain, mechanical

STUDY DESIGN:
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chiropractic Care Only (Active Comparator): 1. The treating clinician will use soft tissue palpation procedures applied to hips, pelvis / buttocks low back and mid back to identify taut and tender regions for manual therapy, e.g., trigger points that the clinician identified during soft tissue palpations.
  2. The treating clinician will use soft tissue treatment procedures, e.g., applying precise pressure to trigger points and manual stretching techniques, to relieve taut and tender regions that were identified during soft tissue palpation procedures.
  3. The treating clinician will perform high velocity, low amplitude (HVLA) spinal adjustments to restricted areas of the mid back, lower back, and hips regions.
  Interventions: Other: Chiropractic Care
- Chiropractic Care Plus Radial Pulse Therapy (Experimental): Chiropractic Care is the same as described for the active comparator arm. After receiving chiropractic care, the subject receives radial extracorporeal shockwave therapy (ESWT). The treating clinician places the ESWT probe over the treatment areas in the mid back, low back, and hip regions. At each clinic visit, there are up to six treatment areas for ESWT. At each treatment area, the subject receives 2000 radial pulses at frequency of 10 Hz (single pulse every 100 ms or 10 pulses per second). The intensity of the radial pulses are comfortable for the subjects. Duration of ESWT at each treatment area is 200 seconds or 3.33 minutes.
  Interventions: Other: Chiropractic Care; Other: Radial Extracorporeal Shockwave Therapy (ESWT) - Radial Pulse Therapy

INTERVENTIONS:
Other: Chiropractic Care — Chiropractic Care is the active comparator arm / intervention. All subjects will receive chiropractic care.
Other: Radial Extracorporeal Shockwave Therapy (ESWT) - Radial Pulse Therapy — This intervention is answering the question: Does on radial ESWT have additive therapeutic effects on the recovery of acute lower back pain symptoms - better or earlier reduction in pain intensity or improvement in physical function - than chiropractic care / manual therapy alone? Subjects will be randomly assigned to receive chiropractic care and ESWT or only chiropractic care.
  Arms: Chiropractic Care Plus Radial Pulse Therapy

SUMMARY:
The goal of this clinical trial is to learn if the addition of radial pulse therapy to chiropractic care will help adult patients recover faster to an acute bout of low back pain. Radial pulse therapy is the application of acoustic waves that passes through the skin to tissues and cells in the body. The main questions that the clinical trial aims to answer are:

* Does the addition of radial pulse therapy to chiropractic care result in better or earlier reduction in pain intensity?
* Does the addition of radial pulse therapy to chiropractic care result in better or earlier improvement in physical function?

Researchers will compare radial pulse therapy plus chiropractic care to chiropractic care alone to see if patients with acute low back pain recover faster with the addition of radial pulse therapy.

Participants will:

* Visit the clinic once a week for 5 weeks
* Receive chiropractic care with or without the addition of radial pulse therapy to the low back and hip regions of the body
* Report their pain intensity and perform a physical function test at each clinic visit

ELIGIBILITY:
Inclusion Criteria:

1. Biological sex of male or female
2. Age Range: 18 to 40 years old
3. Diagnosis of acute mechanical low back pain (< 3 months duration)
4. Pain intensity > 3 on the 11 point NPRS with 0 "being no pain at all" to 10 "being worse pain possible" within the context of either "right now" or "at its worst during the past 7 days"

Exclusion Criteria:

1. Subjects who are currently using over-the-counter nonsteroidal anti-inflammatory drugs (NSAIDs), like ibuprofen (Advil, Motrin) and naproxen (Aleve), or prescription NSAIDs to manage any medical condition.
2. Subjects who used oral corticosteroids that are only available by prescription to manage any medical condition within the past 6 weeks.
3. Subject who received a corticosteroid injection for any medical condition within the past 6 weeks.
4. Subjects who are not willing to be randomly assigned to either of the treatment interventions.
5. Subjects with open wounds to the lower and mid back that will prevent the application of radial ESWT.
6. Subjects with hypermobility and/or instability of the lower and mid back, which are contraindications for manual therapy.
7. Subjects who have a case history of low back pain episodes, e.g., chronic or persistent occurrence of low back pain.
8. Subjects who do not meet the differential diagnosis of acute mechanical low back pain, i.e., origin of their back pain is unknown or non-specific to a low back structure.

   -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity: Numeric Pain Rating Scale (NPRS) | From enrollment to the end of intervention at week 5.
  Before the administration of treatment at each visit, subjects rate their pain on a scale of 0 to 10 with 0 being no pain at all and 10 being worse pain possible. The subjects provide NPRS scores within the context of right now, pain at its best in the past 7 days, and pain at its worst in the past 7 days. At the end of each treatment visit, subjects rate their pain right now on a scale of 0 to 10 with 0 being no pain at all and 10 being worse pain imaginable
Physical Function Assessment of a Squat Test | From enrollment to the end of intervention at week 5.
  1. Before and after the administration of treatment at each visit, subjects perform six squats - moving from a standing position to a squat position. Using an iPad Pro researchers record subjects performing the 3 consecutive squats from a front view and then 3 consecutive squats from a side view. There are 15 seconds between the six squats.
  2. Using the Kinetisense software on the iPad Pro, researchers generate a Clinical Biomechanics Report to measure squat performance.
  3. The overall score from clinical biomechanics report for the squat test is the primary outcome to assess physical function.

SECONDARY OUTCOMES:
Clinical Biomechanics of Squat Performance | From enrollment to the end of intervention at week 5.
  (1) Before and after the administration of treatment at each visit, subjects perform six squats - moving from a standing position to a squat position. Using an iPad Pro researchers record subjects performing the 3 consecutive squats from a front view and then 3 consecutive squats from a side view. There are 15 seconds between the six squats. (2) Using the Kinetisense software on the iPad Pro, researchers generate a Clinical Biomechanics Report to measure squat performance. (3) The secondary outcomes from Clinical Biomechanics Report are: (1) Thighs Reached Horizontal; (2) Knee Valgus; (3) Knee Over Toe; (4) Heels Raised; (5) Shoulder-Wrist Line; (6) Shoulder Lateral Tilt; (7) Shoulder Axis Rotation; and (8) Lumbopelvic Rounding.

CONTACTS AND LOCATIONS:
Locations (1):
- Seneca Falls Health Center at Northeast College of Health Sciences, Seneca Falls, New York, United States

IPD SHARING:
Plan to Share IPD: No